CLINICAL TRIAL: NCT06891794
Title: Use of Cervical Cap and Menstrual Disc for Application of Topical Anesthetic Prior to Intrauterine Device (IUD) Insertion
Brief Title: Use of Cervical Cap and Menstrual Disc for Application of Topical Anesthetic Prior to IUD Insertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Julia Tasset, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OHSU IRB 28118
Record Dates: First submitted 2025-03-06; First posted 2025-03-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: IUD
Keywords: Topical Anesthetic; IUD Insertion
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination; Contraceptive Devices, Female

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two arms (menstrual disc or cervical cap) for eutectic mixture of local anesthetics (EMLA) cream application prior to intrauterine device (IUD) insertion
Masking Description: This is an open label study that involves no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Menstrual disc (Experimental): Participants will be provided with a menstrual disc filled with 5mg of 2.5% prilocaine-2.5% lidocaine cream and manufacturer instructions for placement. Study personnel will leave the room, and participants will undress and attempt to place the disc. The provider will return to the room, make sure the disc is correctly placed, and set a seven minute timer. After the seven minute timer, participants will self-remove the disc or the clinician will remove it and place the intrauterine device (IUD) according to manufacturer technique.
  Interventions: Combination Product: Menstrual disc with EMLA cream
- Cervical cap (Experimental): Participants will be provided with a cervical cap filled with 5mg of 2.5% prilocaine-2.5% lidocaine cream and manufacturer instructions for placement. Study personnel will leave the room, and participants will undress and attempt to place the cap. The provider will return to the room, make sure the cap is correctly placed, and set a seven minute timer. After the seven minute timer, participants will self-remove the cap or the clinician will remove it and place the intrauterine device (IUD) according to manufacturer technique.
  Interventions: Combination Product: Cervical cap with EMLA cream

INTERVENTIONS:
Combination Product: Menstrual disc with EMLA cream — Eutectic mixture of local anesthetics (EMLA) cream self-administered using a menstrual disc
  Other Names: 2.5% prilocaine-2.5% lidocaine cream; Softdisc
  Arms: Menstrual disc
Combination Product: Cervical cap with EMLA cream — Eutectic mixture of local anesthetics (EMLA) cream self-administered using a menstrual disc
  Other Names: FemCap; 2.5% prilocaine-2.5% lidocaine cream
  Arms: Cervical cap

SUMMARY:
This prospective, open label, double arm, feasibility group study will recruit participants planning to undergo office intrauterine device (IUD) placement without sedation or anxiolysis at the Center for Women's Health. Participants will self-administer a topical anesthetic using a contraceptive cervical cap or menstrual disc.

Twenty-four nulliparous women will be recruited to receive one of two administration methods immediately prior to IUD placement (12 subjects in each arm): 1) menstrual disc filled with 5g eutectic mixture of local anesthetics (EMLA) cream or 2) cervical cap filled with 5g EMLA cream.

DETAILED DESCRIPTION:
Nulliparous patients undergoing IUD insertion will administer EMLA cream by menstrual disc or cervical cap prior to insertion. The medical provider will ensure proper placement of the cap or disc and perform a bi-manual exam to assess the patient's uterine position. A seven minute timer will be set, the cap/disc will be removed, and the provider will proceed with the IUD insertion according to manufacturer technique.

Visual Analog Scale (VAS) scores will be used throughout the procedure to assess participant pain throughout insertion. Participants and providers will report on pain, side effects, and procedure complications immediately after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for IUD placement at the Center for Women's Health in Complex Family Planning clinic
* Able to review and sign study consents in English
* Generally healthy

Exclusion Criteria:

* History of any prior births, miscarriages, or abortions after 16 weeks' gestation
* Currently pregnant, known or suspected
* Current stringless IUD in place
* Participants premedicated with misoprostol
* History of chronic pelvic pain which patients take daily medication for
* History of endometriosis, fibroids, adenomyosis, prior cervical procedures (such as Loop Electrosurgical Excision Procedure (LEEP) or cold knife cone)
* Any contraindications to IUD placement (per current labeling including pregnancy, fibroids that distort the uterine cavity, exam consistent with pelvic inflammatory disease, allergy to any component of the levonorgestrel intrauterine system (LNG-IUS), etc.)
* Known allergy to eutectic mixture of local anesthetics (EMLA) or lidocaine cream, silicone, menstrual disc, or cervical cap
* Any contraindication to EMLA or lidocaine cream, menstrual disc, or cervical cap
* Previous IUD placement or failed attempt of an IUD placement
* Weight < 54.4kg (120 lbs)
* Plan for use of oral anxiolysis, moderate/deep sedation, or narcotics for procedure
* Patient requesting or patient use in the past 24 hours of oral anxiolysis, moderate/deep sedation, or narcotics
* Any planned concomitant procedures, such as dilation and curettage (D&C), endometrial biopsy, colposcopy, hysteroscopy, etc.
* Illicit drug use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Successful Placement | Immediately after IUD placement procedure
  The number of participants able to correctly place the cap or disc as instructed, assessed by provider
Satisfaction with pain control | Immediately after IUD placement procedure
  Participant-reported satisfaction with pain control for IUD placement using EMLA cream measured the Patient Acceptable Symptom State (PASS) methodology.

SECONDARY OUTCOMES:
Ease of cap/disc placement | Immediately after IUD placement procedure
  Participant-reported ease of placement of menstrual cap or disc. Response options will be "very easy", "somewhat easy", "neutral", "somewhat difficult", and "very difficult".
Protocol deviations | Immediately after IUD placement procedure
  Provider-reported deviations from the standard protocol including need for additional analgesia, oral pain medication, oral anxiolytic medication, need for cervical dilation, rescheduling with sedation per patient preference, or other.
Ease of IUD placement | Immediately after IUD placement procedure
  Provider-reported ease of IUD placement with response options "usual", "difficult", or "very difficult"
Procedure complications | Immediately after IUD placement procedure
  Provider-reported complications of IUD placement procedure including vagal reaction, perforation, placement failure, allergic reaction, or other.
Typical menstrual pain | On the day of IUD placement procedure prior to cap/disc placement and IUD placement
  Patient-reported 11-point Numerical Rating Scale (NRS) of their menstrual pain where 0 represents no pain and 10 represents the worst possible pain.
Pain during IUD placement procedure | Measured throughout IUD placement procedure immediately before the procedure, during placement of disc/cap, during speculum placement, during tenaculum placement, during sounding, during IUD placement, and 5 minutes after completion
  Patient-reported pain using a 100 millimeter Visual Analog Scale (VAS) throughout IUD placement procedure. Participants will mark their level of pain along a 100mm line, where one end (0) represents no pain and the other represents the worst possible pain (100). The distance from the "no pain" end to the participant's mark is measured to provide a numeric representation of pain
Acceptability of pain mangement | one day post-procedure
  Patient-reported acceptability of pain management measured by a 5-point Likert scale question. Participants will be asked "How would you rate your satisfaction with the pain control during your IUD placement?". Response options range from very satisfied (1) to very dissatisfied (5).

OTHER OUTCOMES:
Reasons for non-participation | During screening/enrollment at the time when an eligible participant declines participation
  For eligible prospective participants who were approached but declined participation, they will be asked the reason why they chose not to participate. This will be an open-ended response where the study staff member performing the screening will record the reason for declining participation.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Tasset, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States